CLINICAL TRIAL: NCT04807322
Title: Reverse Total Shoulder Arthroplasty in Patients Who Exceeded Their Life-expectancy: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Bürgerspital Solothurn (Other)
Responsible Party: Principal Investigator, Mai Lan Dao Trong, Attending physician shoulder and elbow surgery, Bürgerspital Solothurn
Other Study IDs: RTSA in very old patients
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Reverse Total Shoulder Arthroplasty
Keywords: reverse total shoulder arthroplasty; RTSA; elderly; proximal humerus fracture; cuff arthropathy; outcome; complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elective cases: Patients, who received a RTSA for degenerative reasons like cuff arthropathy or osteoarthritis
  Interventions: Procedure: Reverse Total Shoulder Arthroplasty (RTSA)
- Fracture cases: Patients, who received a RTSA for a proximal humerus fracture
  Interventions: Procedure: Reverse Total Shoulder Arthroplasty (RTSA)

INTERVENTIONS:
Procedure: Reverse Total Shoulder Arthroplasty (RTSA) — Implantation of a Reverse Total Shoulder Arthroplasty

SUMMARY:
Reverse total shoulder arthroplasty (RTSA) has become an established treatment for cuff arthropathy, severe osteoarthritis and in certain fracture cases. Due to the increasingly aging population, patients who have already exceeded their life-expectancy pose a significant challenge to the shoulder surgeon. Therefore, we wanted to investigate patient demographics, hospital stay length, complication rate functional outcome, patient reported outcome scores and mortality retrospectively for patients, who were older than 83 years at time of implantation of a RTSA.

DETAILED DESCRIPTION:
This is a retrospective single institution study. All patients older than 83 years who received a reverse shoulder arthroplasty from 2008 until 2019 are included. Elective cases are compared to fracture cases (patient demographics, length of hospital stay, complication rate, functional outcome, patient reported outcome scores and mortality).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 83 years at time of surgery
* Patients who received a reverse total shoulder arthroplasty

Exclusion Criteria:

* Patients younger than 83 years at time of surgery

Min Age: 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients who have already exceeded their life-expectancy (83 years in Switzerland)
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-03-24 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Patient reported outcome score: ASES | until august 2020
  American Shoulder and Elbow Society (ASES) Score
Complication rate | until august 2020
  postoperative complications requiring surgical intervention
Quality adjusted life year (QALY) | until august 2020
  The quality adjusted life year (QALY) ) is a well-established indicator of the life quality for the remaining years and was calculated as the years of life following the operation, multiplied by the utility value, for the current study, defined as the postoperative American Shoulder and Elbow Surgeons Shoulder Score (ASES) score (0-1 points) at last follow-up.
Mortality | until august 2020
  Survivership
Patient reported outcome score: QuickDASH | until august 2020
  Quick Disabilities of the arm, shoulder and hand (DASH) Score,
Patient reported outcome score: VAS | until august 2020
  Visual analog score (VAS)

SECONDARY OUTCOMES:
Patient demographics | at time of surgery
  male/female ratio, age, BMI, ASA (American Society of Anesthesiologists) classification, hospital stay length, range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Mai Lan Dao Trong, MD, Principal Investigator — Bürgerspital Solothurn
Locations (1):
- Bürgerspital Solothurn, Solothurn, Switzerland

IPD SHARING:
Plan to Share IPD: No